CLINICAL TRIAL: NCT02540538
Title: Safety and Immunogenicity of HBAI20 Hepatitis B Vaccine in Naive Adults and Non-responders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: CyTuVax (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HBnr01; 2014-000913-30 (EudraCT Number)
Record Dates: First submitted 2015-08-25; First posted 2015-09-04 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Hepatitis B
Keywords: Adjuvants, immunologic; Interleukin-2; Hepatitis B vaccines; Non-responders
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HB vaccine naive - HBVaxPro (Active Comparator): Subjects have never been vaccinated with a Hepatitis B vaccine. Subjects are vaccinated with Hepatitis B vaccine HBVaxPro-10ug at day 0, 30, and 180.
  Interventions: Biological: HBVaxPro
- HB vaccine naive - HBAI20 (Experimental): Subjects have never been vaccinated with a Hepatitis B vaccine. Subjects are vaccinated with Hepatitis B vaccine HBAI20 at day 0 and 30, and Hepatitis B vaccine HBVaxPro-10ug at day 180.
  Interventions: Biological: HBAI20
- Non-responders - HBAI20 (Experimental): Subjects have been vaccinated 6 times with a Hepatitis B vaccine without developing a protective immune response, measured as anti Hepatitis B surface antigen antibodies, superior to 10mIU/ml.
  Subjects are vaccinated with Hepatitis B vaccine HBAI20 at day 0 and 30, and Hepatitis B vaccine HBVaxPro-10ug at day 180.
  Interventions: Biological: HBAI20

INTERVENTIONS:
Biological: HBVaxPro — 3 vaccinations with HBVaxPro-10ug at 0, 30, and 180 days.
  Arms: HB vaccine naive - HBVaxPro
Biological: HBAI20 — 2 vaccinations with HBAI20 at 0 and 30 days and 1 vaccination with HBVaxPro-10ug at 180 days.
  Arms: HB vaccine naive - HBAI20; Non-responders - HBAI20

SUMMARY:
The purpose of this study is to determine whether the HBAI20 vaccine is safe and more immunogenic than the HBVaxPro-10µg in people who have never been vaccinated with a hepatitis B vaccine and in people who have been vaccinated 6 times with hepatitis B vaccine but do not have a protective anti hepatitis B antibody titer.

DETAILED DESCRIPTION:
Rationale: Worldwide, people are suffering from the consequences of Hepatitis B (HB) virus infection. Currently available vaccines are protective in most of the vaccinees, however, a small part of the population does not respond to these vaccines (non-responders). A new adjuvant (AI20) has been developed by CyTuVax to improve the standard Hepatitis B vaccine for the protection of non-responders. The AI20 adjuvant consists of depot-attached rhuIL-2 (aggregated Interleukin-2 molecules attached to alum), facilitating the slow release of highly concentrated IL-2 nano aggregates. As shown in preclinical experiments, vaccination of mice, rats, and rabbits with the new HBAI20 vaccine results in higher and earlier immune responses to Hepatitis B surface antigen (HBsAg) compared to vaccination with one of the standard Hepatitis B vaccines. This clinical study will be done in order to assess the safety of the AI20 adjuvant and test if the AI20 adjuvanted Hepatitis B vaccine induces protective antibody titers in the vaccinated non-responders.

Objective: In the current study we investigate the safety of the HBAI20 vaccine. Furthermore, the efficacy of the HBAI20 vaccine in non-responders is investigated.

Study design: Partly double blinded randomized controlled intervention phase I study, partly open-label phase I study.

Study population: Healthy volunteers (n=24) and registered non-responders (n=12), 18-59 years old, males and females.

Intervention: The study will include 3 groups. HB vaccine naïve healthy subjects are randomized into group 1 and 2 and registered non-responders are included in group 3.

"Group 1" subjects receive the standard HB vaccine (HBVaxPro-10µg), "Group 2" and "Group 3" subjects receive the HBAI20 vaccine. 2 subjects from "Group 3" will constitute "Group 3 pilot" and will start the study 7 days before the start of the remaining "Group 3" subjects.

All study subjects in groups 2 and 3 will receive two vaccinations with the assigned investigational medical product (IMP) at 0 and 1 month and one regular booster vaccination with the standard HB vaccine HBVaxPro-10µg 6 months after the first dose according to the recommended vaccination schedule for HBVaxPro-10µg.

Main study parameters/endpoints: The primary study parameter is the number and intensity of local and systemic adverse reactions (redness, swelling, impaired movement). The secondary study parameter is the HBAI20 vaccine immunogenicity as calculated by the median titer, geometric mean titer, geometric mean titer increase, proportion of subjects with a virus specific antibody titer measure by the COBAS system of ≥ 10 mIU/ml, and seroconversion rate. Seroconversion is defined as a four-fold increase in titer or a conversion from seronegative to an anti-HBsAg antibody titer of more than 10 mIU/ml after vaccinations.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Study subjects will be vaccinated 3 times at 0, 1 and 6 months from the beginning of the study and invited to the hospital for 8 visits. The risks associated with participation in this study are considered to be low and comparable with standard vaccines. Physical discomfort after vaccine administration can occur at the injection site (redness, swelling, etc.) and systemically (fever, fatigue, headache). Effects are expected to occur for a short period of time (within the first 4 days after the first and second injection). In addition subjects may experience adverse reactions to the cytokine component of the adjuvant. Because of the very low dose of the cytokine component of the adjuvant, which will be gradually released, the risks are expected to be low. The potential risks of venepuncture for blood sampling are mild pain and haematoma, and are considered low.

The naïve subjects participating in this study will benefit from participating by receiving immunization against Hepatitis B. Subjects in the non-responder group may benefit when they become responders due to the effect of the HBAI20 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* In good health as determined by the outcome of medical history, physical examination screening/baseline labs and clinical judgment of the clinical investigator
* Age 18 to 59 years, inclusive at the time of enrolment
* Willing and able to adhere to the study regimen
* Having a signed informed consent form

Non-responders:

- Documented non-responders: Subjects with documented two cycles of Hepatitis B vaccination (total of 6 vaccinations) and titer analysis that show that they have not developed the Hepatitis B antibody titer recommended after standard vaccination: anti-HBsAg antibody titer higher to 10mIU/ml.

Exclusion Criteria:

* Any infectious disease at the time of screening and/or enrolment
* Positive HIV, Hepatitis B virus or Hepatitis C virus serology
* Positive anti-IL-2 antibody titer
* Known or suspected immune deficiency
* Known or suspected disease that influences the immune system including chronic allergies that require frequent anti-allergy medication, cancer and transplantation recipients
* Known or suspected allergy to any of the vaccine components.
* Dialysis patient
* History of unusual or severe reactions to any previous vaccination
* History of any neurologic disorder, including epilepsy and autism
* Use of medication that influences the immune system (immune suppressive treatment)
* Any vaccination within 3 months before screening
* Blood donation within 1 month before screening
* Administration of plasma (incl. immunoglobulins) or blood products within 12 months before screening
* Participation in another clinical trial within 3 months before screening
* Abnormal pre-treatment laboratory parameters which are clinically relevant according to the investigator
* Bleeding disorders, or use of medication for bleeding disorders, and use of anti-coagulants
* Female subjects planning to become pregnant or breastfeeding babies until visit 7
* Females: positive urine pregnancy test. Urine test positive at screening date or positive urine pregnancy test on the day of vaccination
* Excessive alcohol or controlled drug use - More than 2 alcohol measures per day (one alcohol measure is a beer (250ml) or one glass of wine (125ml) or one strong measure (35ml) or one port/sherry (75ml)). Regular use of controlled drugs

Exclusion criterion for Hepatitis B naïve subjects (groups 1 and 2):

- Previous vaccination with Hepatitis B vaccine

Exclusion criterion for non-responders (group 3):

- Any Hepatitis B vaccination in the last 6 months

Temporary exclusion criterion for vaccination

- Ear temperature > 38.4°C will lead to postponement of participation and vaccination. Screening may continue when the temperature has normalized.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid ML Oude Lashof, PhD, MD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

REFERENCES:
- [Result] Koc OM, Savelkoul PHM, van Loo IHM, Peeters A, Oude Lashof AML. Safety and immunogenicity of HBAI20 Hepatitis B vaccine in healthy naive and nonresponding adults. J Viral Hepat. 2018 Sep;25(9):1048-1056. doi: 10.1111/jvh.12909. Epub 2018 May 9. PMID 29660190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase I study involved two trials: a double-blinded RCT in naïve participants and an open-label study in a cohort of true non-responders. At the first visit, a physical examination was performed and blood and urine sampling were taken, and informed written consent was required to participate in the study.
Pre-assignment Details: In RCT, 27 recruits, 3 naïve participants exclusions:
  * 1 with liver LFTs abnormalities
  * 1 with anti-HBs-AB >10 mIU/mL
  * 1 with suspicion of Cushing's syndrome Thus, 24 healthy participants were included.
  In the open-label study, 10 true non-responders were screened, then included. All participants were between 18 and 59 years of age.
Groups:
- Non-responders - HBAI20: Subjects have been vaccinated 6 times with a Hepatitis B vaccine without developing a protective immune response, measured as anti Hepatitis B surface antigen antibodies, superior to 10mIU/ml.
  Subjects are vaccinated with Hepatitis B vaccine HBAI20 at day 0 and 30, and Hepatitis B vaccine HBVaxPro-10ug at day 180.
  HBAI20: 2 vaccinations with HBAI20 at 0 and 30 days and 1 vaccination with HBVaxPro-10ug at 180 days.
Period: Overall Study
Arm/Group | HB Vaccine Naive - HBVaxPro | HB Vaccine Naive - HBAI20 | Non-responders - HBAI20
Started | 12 | 12 | 10
Completed | 12 | 11 | 10
Not Completed | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: RCT: 27 participants screened, 3 excluded: 1 with LFTs abnormalities, 1 anti-HBs titre >10 mIU/mL, 1 suspected Cushing's syndrome. 24 included. Open-Label: 10 screened and included.
Groups:
- Total: Total of all reporting groups
Arm/Group | HB Vaccine Naive - HBVaxPro | HB Vaccine Naive - HBAI20 | Non-responders - HBAI20 | Total
Number analyzed (Participants) | 12 | 12 | 10 | 34
Age, Continuous [Mean (Inter-Quartile Range); unit: Years (IQR)] | 29 [22 to 35] | 29 [22 to 32] | 48 [42 to 58] | 34 [23 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 5 | 22
  Male | 4 | 3 | 5 | 12
BMI [Mean (Inter-Quartile Range); unit: kg/m^2] | 25 [20 to 25] | 23 [22 to 27] | 29 [24 to 31] | 25 [22 to 29]
Anti-HBs Titers < 2 IU/ml [Count of Participants; unit: Participants] — Number of participants with Anti-HBs titers lower than 2 IU/ml
  Participants | 12 | 12 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Local and/or General Adverse Events Irrespective of Severity
Description: Subjects will be given a diary for 4 days after the first and second vaccination.
  Dairy: Local reactions at injection site: Pain (1 to 4), Impaired movement of injected arm (1 to 4), Redness/erythema (cm), Swelling (cm), Induration (cm) General/Systemic adverse events: Fever (temperature measurement), Headache (1 to 4), Fatigue (1 to 4), Muscle pain (1 to 4), Skin rash (1 to 4), Vomiting (1 to 4), Diarrhea (1 to 4).
  Record medication taken during the study (up to 7 months after the first vaccination).
Time Frame: Up to 7 months after first vaccination.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HB Vaccine Naive - HBVaxPro | HB Vaccine Naive - HBAI20 | Non-responders - HBAI20
Number analyzed (Participants) | 12 | 12 | 10
Participants
  Pain at the injection site | 8 | 9 | 7
  Impaired movement of injected arm | 7 | 8 | 4
  Redness/Erythema | 6 | 4 | 4
  Swelling | 3 | 2 | 0
  Induration | 1 | 1 | 4
  Fever | 0 | 0 | 1
  Headache | 4 | 3 | 1
  Fatigue | 5 | 3 | 3
  Myalgia | 9 | 9 | 7
  Vomiting | 0 | 1 | 0
  Diarrhea | 2 | 3 | 0

2. Primary Outcome: Subjects With Local and/or General SEVERE Adverse Events
Description: Subjects will be given a diary for 4 days after the first and second vaccination.
  Dairy: Local reactions at injection site: Pain (1 to 4), Impaired movement of injected arm (1 to 4), Redness/erythema (cm), Swelling (cm), Induration (cm) General/Systemic adverse events: Fever (temperature measurement), Headache (1 to 4), Fatigue (1 to 4), Muscle pain (1 to 4), Skin rash (1 to 4), Vomiting (1 to 4), Diarrhea (1 to 4).
  Record medication taken during the study (up to 7 months after the first vaccination).
  The laboratory parameters analysed at day 10, 30, 40, 60, 180, and 210 are:
  Hematology: Hematocrit, Hemoglobin, RBC count, WBC count, Platelet count, Neutrophils, Eosinophils, Basophils, Lymphocytes, and Monocytes. Biochemistry: Creatinine, Albumin, Alkaline Phosphatase, Total Bilirubin, ALT (GPT), AST (GOT), Gamma-Gt, C-Reactive Protein, and TSH/FT4.
  Urinalysis (day 10, 40, and 210): Clarity, Color, Specific gravity, Leukocytes, Nitrite, pH, Erythrocytes, Albumin, and Glucose.
Time Frame: Up to 7 months after first vaccination
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HB Vaccine Naive - HBVaxPro | HB Vaccine Naive - HBAI20 | Non-responders - HBAI20
Number analyzed (Participants) | 12 | 12 | 10
Participants
  Severe pain at injection site | 0 | 0 | 0
  Severe impaired movement of injected arm | 0 | 0 | 0
  Severe redness | 1 | 0 | 1
  Sever swelling | 0 | 0 | 0
  Severe induration | 0 | 0 | 1
  Fever | 0 | 0 | 0
  Headache | 0 | 1 | 0
  Fatigue | 0 | 0 | 0
  Myalgia | 0 | 0 | 0
  Vomiting | 0 | 0 | 0
  Diarrhea | 0 | 1 | 0

3. Secondary Outcome: Number of Participants With Seroprotection
Description: Seroprotection at visit number 7, one month after the third vaccination. Anti-HBs antibodies were assayed from serum using a routine chemiluminescence assay (Anti-HBs, Cobas 8000, Roche, Germany). Titres >10 mIU/mL were considered to be seroprotective.
Time Frame: Day 0, 10, 30, 40, 60, 180, and 210
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HB Vaccine Naive - HBVaxPro | HB Vaccine Naive - HBAI20 | Non-responders - HBAI20
Number analyzed (Participants) | 12 | 12 | 10
Participants
  Day 10 | 0 | 0 | 3
  Day 30 | 1 | 2 | 1
  Day 40 | 7 | 11 | 6
  Day 60 | 9 | 10 | 6
  Day 180 | 10 | 9 | 7
  Day 210 | 12 | 12 | 9

ADVERSE EVENTS:
Time Frame: Up to 7 months after first vaccination
Arm/Group | HB Vaccine Naive - HBVaxPro | HB Vaccine Naive - HBAI20 | Non-responders - HBAI20
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 2/12 | 4/12 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HB Vaccine Naive - HBVaxPro (N=12) | HB Vaccine Naive - HBAI20 (N=12) | Non-responders - HBAI20 (N=10)
Unsolicited symptoms (General disorders) | 2 | 4 | 5

LIMITATIONS AND CAVEATS:
We are aware of the limitations of the small study population when drawing the tentative conclusions from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No